CLINICAL TRIAL: NCT03632642
Title: Pilot Randomised Controlled Trial of Penicillin Versus Flucloxacillin for Definitive Treatment of Invasive Penicillin Susceptible Staphylococcus Aureus
Brief Title: Penicillin Against Flucloxacillin Treatment Evaluation
Acronym: PANFLUTE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never commenced
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREC/17/QRBW/620
Record Dates: First submitted 2018-07-22; First posted 2018-08-15 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2018-08

CONDITIONS: Staphylococcus Aureus
MeSH Terms: conditions — Staphylococcal Infections | interventions — Penicillin G; Floxacillin

STUDY DESIGN:
Intervention Model Description: The study will be a pilot open-label multicentre randomised trial that is investigator-initiated comparing two drug regimens: benzylpenicillin vs. flucloxacillin for penicillin susceptible S. aureus bloodstream infections. We will aim to enrol 60 patients (30 in each arm) over a 12-month period. The participation duration for each enrolled patient is 90 days. Data will be collected for the participants from the date of when the first positive blood culture was obtained, which will be within 72 hours of enrollment. Consented patients will be randomised on day 1 (the day of randomisation) to either benzylpenicillin or flucloxacillin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Benzylpenicillin arm (Active Comparator): Patients randomised to benzylpenicillin will be treated according to Therapeutic Guidelines 15th Edition. During hospitalisation, the standard dose will be 1.8g Q4H IVI for uncomplicated BSIs and 2.4g Q4H for deep-seated or critical illness infections.
  Interventions: Drug: Benzylpenicillin
- Flucloxacillin arm (Active Comparator): Patients randomised to flucloxacillin will be treated according to Therapeutic Guidelines 15th Edition. During hospitalisation, the standard dose will be 2g Q6H IVI or 2g Q4H for deep-seated or criticial illness infections.
  Interventions: Drug: Flucloxacillin

INTERVENTIONS:
Drug: Benzylpenicillin — The study drug will be administered for a minimum of 2 weeks (the minimal currently accepted duration of IV therapy for SAB.) For patients who do not fulfill criteria for 2 weeks of therapy, the duration of treatment will be 4 to 6 weeks and will be made by the treating clinician.
  Arms: Benzylpenicillin arm
Drug: Flucloxacillin — The study drug will be administered for a minimum of 2 weeks (the minimal currently accepted duration of IV therapy for SAB.) For patients who do not fulfill criteria for 2 weeks of therapy, the duration of treatment will be 4 to 6 weeks and will be made by the treating clinician.
  Arms: Flucloxacillin arm

SUMMARY:
There is theroretical superiority with benzylpenicillin over orther anti-staphylococcal penicillins (ASP) for treatment of penicillin susceptible S. aureus (PSSA) infections due to a lower MIC distribution when compared with ASPs active against PSSA, combined with the ability to obtain higher levels of free non-protein-bound plasma drug concentrations. Although the data to support this theoretical advantage is limited, many clinicians in Australia (and worldwide) use benzylpenicillin for therapy in this situation despite many international guidelines cautioning against this. This uncertainty is significant given that 1) S. aureus bacteraemia (SAB) is associated with a high mortality and significant morbidity, 2) S. aureus is one of the most common organisms isolated from blood cultures, 3) SAB is the most common reason for consultation with an Infectious Disease specialist (which itself has been shown to improve outcomes) and 4) a significant proportion (up to 20%) of SAB isolates in Australia will be reported as susceptible to penicillin, a proportion which appears to be increasing over the past 10 years in Australia and internationally.

Given the frequency of PSSA and the associated morbidity and mortality related to SABs in general, a definitive study to determine the optimal therapy for PSSA is required. In a recent survey of Infectious Diseases Physicians and Clinical Microbiologists in Australasia, 87% of respondents were willing to randomise patients to either benzylpenicillin or flucloxacillin for a clinical trial, whist 71% responded that they would switch therapy from flucloxacillin to benzylpenicillin for treatment of PSSA BSIs in clinical practice (unpublished data).

Therefore, the investigators see the opportunity to determine the feasibility of a definitive study comparing benzylpenicillin against flucloxacillin (or other ASP) for treatment of PSSA bloodstream infections.

DETAILED DESCRIPTION:
Background and rationale:

Resistance to penicillin was discovered in Staphylococcus aureus in the mid-1940s, soon after the introduction of penicillin as a therapeutic agent into clinical practice. The emergence of penicillin resistant S. aureus (PRSA) was widely encountered in hospitals thereafter, with some reports finding rates of PRSA rising from 14% to 38% in less than 1 year. Two mechanisms are known that result in resistance to penicillin in staphylococci. The most common, and earliest described, was by the production of a serine β-lactamase, known as penicillinase (PC1), which hydrolyses the β-lactam ring resulting in the production of penicilloic acid. A second mechanism leads to resistance to penicillin and other beta-lactam agents by production of penicillin-binding protein, PBP2a, encoded by mecA. Following the emergence of PRSA, a new class of anti-staphylococcal penicillins were developed that were resistant to hydrolysis of the beta-lactam ring by penicillinase. The isoxazolyl-penicillins, semi-synthetic penicillin derivatives that are stable during exposure to penicillinase, are now the most commonly used agents for the treatment of S. aureus infections.

Despite widespread resistance to penicillin amongst S. aureus, a significant proportion of invasive isolates remain susceptible. Although penicillin and isoxazolyl-penicillins have been used in clinical practice for more than 50 years, the optimal therapy for patients with invasive penicillin susceptible S. aureus (PSSA) remains controversial. Methicillin susceptible S. aureus (MSSA) bloodstream infections are commonly sub-divided into categories based upon the presence of penicillinase, the absence of which defines PSSA strains. Many clinicians advocate treating both MSSA and PSSA the same, irrespective of whether penicillinase is detected or not. One group who strongly supports this view is the American Heart Association, which has published recently updated guidelines on infective endocarditis. This recommendation is based upon literature suggesting that detection of penicillinase is not reliable in some clinical laboratories. Multiple publications have demonstrated that the previous widely used phenotypic method of penicillinase detection, by nitrocefin hydrolysis, lacks adequate sensitivity for detecting penicillinase. Yet, treatment failure with penicillin due to inability to detect penicillinase has not been previously described in the medical literature to our knowledge. Regardless, many laboratories have now changed methods to the penicillin disc test, where isolates harbouring penicillinase may be detected by interrogation of the edge of the disc, with a sharp edge confirming the presence of penicillinase and a tapered edge indicating an absence. This method is now employed in most Pathology services and is the method approved by international governance organisations.

Other experts argue for potential superiority with penicillin due to a lower MIC distribution when compared with other beta-lactam agents active against S. aureus, combined with the ability to obtain high levels of free non-protein-bound plasma drug concentrations.

To date there is only one previous study that has directly compared the outcome between a semi-synthetic penicillin derivative (dicloxacillin) and penicillin for PSSA infections. In this retrospective study, no statistically significant difference was observed between penicillin and dicloxacillin based on a mortality outcome. Although this study does not support improved outcome with penicillin compared with dicloxacillin, it should be noted that significantly more patients treated with penicillin had a higher Pitt bacteraemia score and deep-seated infection such as endocarditis or osteomyelitis. Data from the ANZCOSS study, a prospective observational study of SAB within Australia between 2007 - 2016, demonstrated a possible 30-day crude mortality benefit for patients treated with benzylpenicillin compared to flucloxacillin or dicloxacillin (unpublished data). Patients in this cohort were treated 2:1 with flucloxacillin over benzylpenicillin, however, benzylpenicillin treatment was proportionally higher in patients with endocarditis or other deep-seated infections. In a multivariate logistic regression model, Flucloxacillin therapy was associated with a non-statistically significant increase in the odds ratio for 30-day mortality (OR 1.55, 95% CI 0.99 - 2.47).

A number of recent studies internationally have reported a resurgence of PSSA, and in particular within the Australian setting, it was noted that 20% of S. aureus bacteraemias (SAB) were found to be susceptible to penicillin in 2013. Given the resurgence of PSSA and the associated morbidity and mortality related to SABs in general, a definitive study to determine the optimal therapy for PSSA is required.

A pilot randomised controlled trial is critical to determining the feasibility for a definitive study due to PSSA BSIs and in order to calculate an appropriate sample size based upon the proportion of deep-seated infections. A definitive trial would greatly enhance the medical literature and help to define the optimum treatment which for both penicillin susceptible and penicillin non-susceptible MSSA in invasive infections, at present, remains unclear.

Objectives and hypothesis:

The investigators hypothesise that penicillin is superior to flucloxacillin for treatment of penicillin susceptible S. aureus bloodstream infections based upon a lower distribution of MICs for penicillin, a higher level of free non-protein-bound drug concentration and favourable side effect profile.

Primary objective:

1. To determine feasibility of a randomised controlled trial of penicillin versus flucloxacillin for definitive management of penicillin susceptible S. aureus bacteraemia

Secondary objective:

1. To assist in calculating an appropriate sample size for a definitive study
2. To determine the proportion of deep-seated infections
3. To determine the feasibility of desirability of outcome rankings (DOOR) as a clinical endpoint

Study design:

The study will be a pilot open-label multicentre randomised trial that is investigator-initiated comparing two drug regimens: benzylpenicillin vs. flucloxacillin for penicillin susceptible S. aureus bloodstream infections. The investigators will aim to enroll 60 patients over a 24-month period. The participation duration for each enrolled patient is 90 days. Data will be collected for the participants from the date of when the first positive blood culture was obtained, which will be within 72 hours of enrolment.

Consented patients will be randomised on day 1 (the day of randomisation) to either benzylpenicillin or flucloxacillin. Data will be obtained from the medical records (electronic or paper) of each participant. Data collected will include relevant investigations (FBC, ELFT, blood culture results, and CRP), any SAE that have occurred, antibiotics administered and evidence of relapse or treatment failure. Participants who are discharged will be followed weekly in outpatients for the duration of intravenous therapy. Participants will be reviewed at day 90 in outpatient clinic if they have been discharged (or within 1-2 weeks thereafter). For participants who do not attend the outpatients clinic, contact will be made by telephone. If attempts at contact are unsuccessful, then the site investigator will review the medical records of the participants at 6-month time intervals until either the vital status has been completed or the study period is complete.

Intervention Participants will be randomised to either benzylpencillin or flucloxacillin. Dosage, frequency and duration of antibiotics will be determined by the treating clinician based upon national guidelines, eTG (Therapeutic Guidelines 15th Edition) as summarised below.

The study drug will be administered for a minimum of 2 weeks (the minimal currently accepted duration of IV therapy for SAB.) Participants treated for 2 weeks will have to meet the following criteria:

* Negative BC at 48-72 hours from first effective antibiotics
* Rapid resolution of fever
* Normal valvular morphology and no evidence of valvular lesions on TTE or TOE
* An identifiable source of infection that has been removed, including drainage of simple skin infections
* No evidence of metastatic focus
* No intravascular prosthetic material
* No significant immunocompromise including any congenital or acquired quantitative or qualitative deficiency of phagocytic cells, complement, or humoral or cell-mediated immunity. This includes:

  * Stem cell or organ transplant recipient
  * Absolute neutrophil count less than 500/μl
  * HIV
  * Prednisolone > 25mg/kg/day for 1 month or cumulative dose > 700mg within 3 months of onset of SAB
  * Use of a monoclonal antibody within 1 month of SAB onset For participants who do not fulfil these criteria, the duration of treatment will be 4 to 6 weeks and will be made by the treating clinician.

Other antimicrobials active against S. aureus will be discouraged during the duration of IV therapy:

Any missed doses of antibiotics will be recorded on the CRF. In order to ensure equivalence amongst the sites, TDM will not be employed during the study for the purpose of tailored antibiotic dosing. Therefore, to ensure participants are treated optimally, dosing will be based upon standard uncomplicated BSIs or critical illness/deep-seated infection and dosed as per eTG. Participants who were initially stratified as uncomplicated BSI may be changed to deep-seated or critical illness if the participants fulfil the criteria after enrolment.

For participants with obesity or renal impairment, dosing may follow local guidelines. All outpatient therapy will be administered by continuous intravenous infusion (CIV). CIV will be discouraged for inpatients, however, if the treating clinician considers this to be necessary, then it will be allowed and recorded in the CRF. Non-antibiotic related management of the participants will be at the discretion of the treating clinician.

Dosing in renal impairment:

Flucloxacillin

* Standard Dose: 2g Q6H (8g/24 hours CIV if home IV therapy)
* Critical Illness or Deep-seated infection: 2g Q4H (12g/24 hours CIV if home IV therapy)
* CrCl <50 ml/min and > 10 ml/min: No change to dose
* CrCl <10 ml/min or on haemodialysis: 50% reduction of dose
* On continuous renal replacement therapy: 2g Q6H

Benzylpenicillin

* Standard Dose: 1.8g Q4H (10.8g/24 hours CIV if home IV therapy)
* Critical Illness or Deep-seated infection: 2.4g Q4H (14.4g/24 hours CIV if home IV therapy)
* CrCl <50 ml/min and > 10 ml/min: 25% reduction of dose
* CrCl <10 ml/min or on haemodialysis: 50% reduction of dose
* On continuous renal replacement therapy:1.8g Q4H

Change of therapy:

Any change to the intervention drug will be discouraged, but left to the discretion of the treating clinician. If an intervention drug needs to be changed (such as due to an adverse event ie. rash) during the intravenous phase of therapy, then this will be a protocol violation. The participant will still remain in the study and be analysed to the group they were randomised, but will be excluded from the per-protocol analysis if the change occurred within the first two weeks from enrolment.

Use of antibiotics with activity against S. aureus after randomisation:

The use of any other antibiotic with activity against S. aureus after randomisation will be discouraged during the intravenous phase of the trial. If a participant requires additional antibiotics due to an indication for broadening antibiotic therapy, the PI should recommend an agent without useful activity towards S. aureus (such as gentamicin, ceftazidime or aztreonam). If a patient receives an antibiotic with activity against S. aureus during the first two weeks of the intravenous phase of the study, this will be recorded as a protocol violation. The participant will still remain in the study and be analysed to the group they were randomised, but will be excluded from the per-protocol analysis. If the participant receives anti-staphylococcal therapy after the first two weeks from enrolment and is still on intravenous therapy with the study drug, they will be included in the per-protocol population. For patients that have completed their intravenous therapy phase of the study but have an indication for ongoing oral therapy, any oral antibiotic may be prescribed and will be recorded in the CRF. The choice of antibiotic and indication for oral therapy is at the discretion of the treating clinician or PI.

Strategies to improve adherence to protocol:

All site PIs will be trained in the study protocol, SOPs and their reporting requirements by the project manager, a study chief investigator or delegate, prior to the site being opened for recruitment. All site PIs will complete a computer-based training course in Good Clinical Practice.

A sticker will be placed in the patient's medical record (one on the progress notes on the day of randomisation, and one in the front inside cover of the medical record if one exists). This sticker will alert clinicians that the patient has been randomised to the PANFLUTE study, with a brief explanation of the study, and confirmation that the participant (or the person responsible) has provided written informed consent.

A copy of the study synopsis will be placed in the bedside chart (observations and drug chart) of the patient. A checklist of study procedures will also be placed in the bedside chart. For sites with electronic medical records and/or prescribing, an electronic "sticker" will be used, and appropriate annotations will be made to the electronic drug chart.

The medication chart (be it paper or electronic) will be checked regularly by the site PI or their delegate (registrar or research nurse) whilst the participant is an inpatient to ensure adherence to the study protocol.

Sample Size:

Recruitment will be from any adult patient admitted to the study site hospital with a bloodstream infection due to PSSA. Based upon previous retrospective case-control studies, the mortality from S. aureus BSI ranges from 10-30%. A sample size of 60 was chosen based upon feasibility of recruiting participants within the time frame for this pilot study from a total of 8 sites.

Assignment of Intervention:

Participants will be randomised to either of the two arms in a 1:1 ratio using a web based interactive randomisation system. Randomisation will be stratified by site. The randomised sequence allocation will be held on a secure server and not accessible by any investigators of members of study staff. The person enrolling the patient will, following obtaining written informed consent, obtain the treatment allocation by logging onto the web-based database and will then assign the allocated treatment to the patient. As the study will be an open-label design, the site investigators will not be blinded to the intervention, however, the investigators assessing the primary outcome will be.

Outcome Measurement:

This study aims to determine the feasibility of Desirability of Outcome Ranking (DOOR) as a novel outcome method for outcome analysis in clinical trials. Participants are classified according to outcomes by using ordinal categories with the aim to evaluate if an intervention is superior to standard care strategy. This approach takes into account a risk/benefit assessment by including participant centered outcomes such as treatment failure, adverse events and complications of the disease process.

Participants will be ranked according to the following stratification:

1. Alive, Treatment failure or Infectious complication - No, Grade 2 or greater AE - No
2. Alive, Treatment failure or Infectious complication - No, Grade 2 or greater AE - Yes
3. Alive, Treatment failure or Infectious complication - Yes, Grade 2 or greater AE - No
4. Alive, Treatment failure or Infectious complication - Yes, Grade 2 or greater AE - Yes
5. Dead, Treatment failure or Infectious complication - Any, Grade 2 or greater AE - Any

Definitions of DOOR components:

Alive: 90 day status

Treatment Failure (Any one of the following):

* Relapse - Positive blood culture following at least 72 hours after a preceding negative culture
* Persistence - Bacteraemia at day 7 or beyond post randomisation
* Readmission - Readmission to hospital attributable to PSSA infection

Infection complications (Any one of the following):

* Positive sterile site culture (excluding bloodstream) at least 7 days after randomisation
* Positive culture from a new sterile site 48 hours or later after randomisation
* Septic shock or ICU admission 24 hours or later after randomization
* New metastatic event that was not present at randomization and occurs 48 hours or later after randomization

Adverse Events:

Hepatotoxicity (defined according to the Common Terminology Criteria for Adverse Events, version 4.0)

* Grade 1: ULN to 3x ULN of GGT/ALP or AST
* Grade 2: >3 to 5x ULN of GGT/ALP or AST
* Grade 3: 5 to 20x ULN of GGT/ALP or AST
* Grade 4: >20x ULN of GGT/ALP or AST
* Patients with pre-existing abnormal liver function tests:

For patients with pre-existing abnormal liver function tests, hepatotoxicity will still be assessed but will include a greater than 2x rise compared to initial GGT/ALT or AST

Kidney Injury (defined according to the Common Terminology Criteria for Adverse Events, version 4.0)

* Grade 1: Creatinine > 1.5 to 2x baseline and < 350 μmol/L
* Grade 2: Creatinine > 2 to 3x baseline and < 350 μmol/L
* Grade 3: Creatinine > 3x baseline and/or > 350 μmol/L
* Grade 4: Dialysis (if previously not on dialysis)

Phlebitis (Assess according to Visual Infusion Phlebitis Score)

* Grade 1: NA
* Grade 2: VIP score of 1 (Pain but no associated erythema and not requiring a change of IVC or central line)
* Grade 3: VIP score of 2,3 or 4 (Pain, redness and swelling +/- palpable venous cord requiring change of IVC or central line)
* Grade 4: VIP score of 5 (As above but with fever attributable to phlebitis)

Haematologic (Any of the following as defined according to the Common Terminology Criteria for Adverse Events, version 4.0)

Platelets

* Grade 1: LLN - 75 x 10^9
* Grade 2: <75 - 50 x 10^9
* Grade 3: <50 - 25 x 10^9
* Grade 4: < 25 x 10^9

Neutrophil

* Grade 1: LLN - 1.5 x 10^9
* Grade 2: <1.5 - 1.0 x 10^9
* Grade 3: <1 - 0.5 x 10^9
* Grade 4: <0.5 x 10^9

Endpoint Assessment:

The primary endpoint will be assessed by a blinded adjudication committee in order to rank participants according to the DOOR outcomes. This committee will include 2 independent Infectious Diseases Physicians appointed by the trial management committee. The information provided to the committee will not include any participant identifiers or any antibiotic details. The data provided will include:

1. Demographic details (such as age and sex)
2. Comorbidities
3. Clinical details (including focus of infection and relevant investigation results)
4. Date and result of all blood cultures taken during days 1-90
5. Date and result of all other available clinical cultures taken from days 1-90 (e.g., cultures of aspirated pleural fluid or pus).
6. Any adverse events recorded
7. Vital status at day 90 and date of death if applicable.

Additional information will be provided to the adjudication committee providing it does not contain antibiotic data or patient identifiers. Each of the committee members will independently rank participants according to DOOR outcomes. If there is discrepancy between the assessments, the committee will refer to a third independent assessor and the majority will determine the rankings.

Discontinuation/withdrawal of participants from trial treatment:

The participants or NOK have the right to choose to withdraw from the study at any time and the investigator may discontinue a participant from the study or from treatment if deemed appropriate at any time. Reasons why a participant may be withdrawn from the study include, but are not limited to, participant or person responsible request, primary treating clinician's request, participant was enrolled and is ineligible (either arising during the study or was overlooked at time of screening and enrolment). Participants will not be withdrawn due to adverse events, unless the adverse event is life threatening. The decision to withdraw a participant from the study must be discussed with the coordinating investigators.

If the participant or person responsible withdraws consent from participating in the study and also withdraws consent for collection of future information, no further evaluations will be performed, and no additional data will be collected. The sponsors may retain and continue to use any data or samples collected before such withdrawal of consent. Participants that abscond will continue to be followed, if possible, until the end of the trial to avoid missing data. Participants withdrawn from the treatment by the treating clinicians will continue to be followed up to the end of the trial to avoid missing data and will be used in the intention-to-treat analysis. Withdrawn participants will not be replaced. If a participant is withdrawn the reason will be recorded in the database.

Statistical Analysis Plan:

Data for this study will be reported as per CONSORT guidelines. All-cause mortality will be represented in a Kaplan-Meier graph. The primary analysis will be performed by a modified intention to treat principle, whereby all participants with data available for the endpoint will be assessed. A per-protocol analysis will also be performed, whereby participants in this population will have to have received at least 2 weeks of the intravenous phase of the study drug and 90 day outcome data.

A summary of baseline participant characteristics with totals and proportions (%) for categorical variables, and minimum, maximum, inter-quartile ranges and standard deviations for continuous variables will be presented. For assessment of the primary outcome, 2 independent clinicians, blinded to the therapy given to each participant, will assess all participants and rank each participant's outcome according to the pre-designed DOOR groups. The probability that a randomly selected patient will have a better DOOR if assigned to the benzylpenicillin arm vs. the flucloxacillin arm will be estimated along with a confidence interval. If there is no difference in DOOR distributions between the 2 arms, then the probability will be near 50%.

ELIGIBILITY:
Inclusion Criteria:

* Bloodstream infection with Staphylococcus aureus susceptible to penicillin and negative for penicillinase by phenotypic methods.
* No more than 72 hours has elapsed since the first positive blood culture was drawn
* Patient is aged 18 years and over
* The patient or approved proxy is able to provide informed consent

Exclusion Criteria:

* Patient with a recorded allergy to penicillin including:

  1. Hypersensitivity type reaction
  2. Stephens-Johnson syndrome
  3. Rash
  4. Urticaria
* Contraindications based upon other recorded allergies, such as gastrointestinal upset, will be at the discretion of the treating clinician
* Patient with significant polymicrobial bacteraemia (skin contaminants excepted)
* Treated with non-curative intent
* Pregnancy or breast-feeding
* Patient currently receiving concomitant antimicrobials with activity against S. aureus which cannot be ceased or substituted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of DOOR | 90 day
  The primary outcome of the study will utilise a desirability of outcome ranking (DOOR) to assess superiority of benzylpenicillin against flucloxacillin.

SECONDARY OUTCOMES:
Adverse Events | 90 day
  All adverse events
Mortality | 14, 42 and 90 days
  All cause mortality at days 14, 42 and 90
Time to defervescence | From randomisation to any period where a temperature is < 37.5 degrees celsius for greater than or equal to 24 hours
  Defined as either the time from randomisation to a temperature < 37.5 degrees celsius for greater than or equal to 24 hours
Persistent bacteraemia | Day 3 and day 7
  At day 3 and day 7 post randomisation
Microbiologic relapse | Any period within 90 days from randomisation following a negative blood culture at least 3 days prior
  Positive blood culture following at least 72 hours after a preceeding negative culture
Microbiologic treatment failure | Any period within day 14 to day 90 from randomisation
  Positive sterile site culture at least 14 days after randomisation
Healthcare costs | 90 day
  Direct healthcare costs

CONTACTS AND LOCATIONS:
Overall Officials: David Paterson, Principal Investigator — UQCCR
Locations (1):
- Brisbane Private Hospital, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided
As this study is a feasibility pilot study of a planned definitive RCT, it is likely that IPD will be made available to future potential collaborators on a definitive study in order to determine the feasibility, calculate an appropriate sample size and determine if any changes are required to the study protocol and SAP in particular.

REFERENCES:
- [Background] Kirby WM. EXTRACTION OF A HIGHLY POTENT PENICILLIN INACTIVATOR FROM PENICILLIN RESISTANT STAPHYLOCOCCI. Science. 1944 Jun 2;99(2579):452-3. doi: 10.1126/science.99.2579.452. PMID 17798398
- [Background] Baddour LM, Wilson WR, Bayer AS, Fowler VG Jr, Tleyjeh IM, Rybak MJ, Barsic B, Lockhart PB, Gewitz MH, Levison ME, Bolger AF, Steckelberg JM, Baltimore RS, Fink AM, O'Gara P, Taubert KA; American Heart Association Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease of the Council on Cardiovascular Disease in the Young, Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and Stroke Council. Infective Endocarditis in Adults: Diagnosis, Antimicrobial Therapy, and Management of Complications: A Scientific Statement for Healthcare Professionals From the American Heart Association. Circulation. 2015 Oct 13;132(15):1435-86. doi: 10.1161/CIR.0000000000000296. Epub 2015 Sep 15. PMID 26373316
- [Background] Gill VJ, Manning CB, Ingalls CM. Correlation of penicillin minimum inhibitory concentrations and penicillin zone edge appearance with staphylococcal beta-lactamase production. J Clin Microbiol. 1981 Oct;14(4):437-40. doi: 10.1128/jcm.14.4.437-440.1981. PMID 6974738
- [Background] Kaase M, Lenga S, Friedrich S, Szabados F, Sakinc T, Kleine B, Gatermann SG. Comparison of phenotypic methods for penicillinase detection in Staphylococcus aureus. Clin Microbiol Infect. 2008 Jun;14(6):614-6. doi: 10.1111/j.1469-0691.2008.01997.x. Epub 2008 Apr 5. PMID 18397333
- [Background] Coombs GW, Daly DA, Pearson JC, Nimmo GR, Collignon PJ, McLaws ML, Robinson JO, Turnidge JD; Australian Group on Antimicrobial Resistance. Community-onset Staphylococcus aureus Surveillance Programme annual report, 2012. Commun Dis Intell Q Rep. 2014 Mar 31;38(1):E59-69. doi: 10.33321/cdi.2014.38.12. PMID 25409357
- [Background] Nissen JL, Skov R, Knudsen JD, Ostergaard C, Schonheyder HC, Frimodt-Moller N, Benfield T. Effectiveness of penicillin, dicloxacillin and cefuroxime for penicillin-susceptible Staphylococcus aureus bacteraemia: a retrospective, propensity-score-adjusted case-control and cohort analysis. J Antimicrob Chemother. 2013 Aug;68(8):1894-900. doi: 10.1093/jac/dkt108. Epub 2013 Apr 18. PMID 23599360
- [Background] Coombs GW, Daley DA, Thin Lee Y, Pearson JC, Robinson JO, Nimmo GR, Collignon P, Howden BP, Bell JM, Turnidge JD; Australian Group on Antimicrobial Resistance. Australian Group on Antimicrobial Resistance Australian Staphylococcus aureus Sepsis Outcome Programme annual report, 2014. Commun Dis Intell Q Rep. 2016 Jun 30;40(2):E244-54. doi: 10.33321/cdi.2016.40.20. PMID 27522136
- [Background] Cheng MP, Rene P, Cheng AP, Lee TC. Back to the Future: Penicillin-Susceptible Staphylococcus aureus. Am J Med. 2016 Dec;129(12):1331-1333. doi: 10.1016/j.amjmed.2016.01.048. Epub 2016 Feb 26. PMID 26924388
- [Background] Evans SR, Rubin D, Follmann D, Pennello G, Huskins WC, Powers JH, Schoenfeld D, Chuang-Stein C, Cosgrove SE, Fowler VG Jr, Lautenbach E, Chambers HF. Desirability of Outcome Ranking (DOOR) and Response Adjusted for Duration of Antibiotic Risk (RADAR). Clin Infect Dis. 2015 Sep 1;61(5):800-6. doi: 10.1093/cid/civ495. Epub 2015 Jun 25. PMID 26113652